CLINICAL TRIAL: NCT00200447
Title: Assessment of Carbidopa/l-Dopa and Carbidopa/l Dopa/Entacapone on Synaptic Dopamine in Parkinson's Patients: An Open-Label Feasibility/Pilot Study With [123I]-IBZM SPECT (DOPA-SYN)
Brief Title: An Open-Label Feasibility/Pilot Study With [123I]-IBZM SPECT (DOPA-SYN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Molecular NeuroImaging (Other)
Responsible Party: John Seibyl M.D., molecular NeuroImaging
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MNI 0011
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson; brain imaging
MeSH Terms: conditions — Parkinson Disease | interventions — Stalevo

INTERVENTIONS:
Drug: carbidopa/l-dopa
Drug: carbidopa/l-dopa/entacapone
Drug: Stalevo
Procedure: [123I]-IBZM imaging

SUMMARY:
This study conducted to more fully evaluate the way that carbidopa/levodopa and entacapone may work in the brain. This research study uses [123I]-IBZM and dynamic SPECT imaging to determine the amount and the duration of dopamine release from specific regions in the brain after treatment with either the combination of carbidopa/levodopa or the combination of carbidopa/levodopa/entacapone.

DETAILED DESCRIPTION:
This is a pilot evaluation of dopaminergic function in PD using a bolus plus constant infusion protocol with [123I]-IBZM and SPECT to evaluate the potential for carbidopa/l-dopa alone or carbidopa/l-dopa/entacapone to produce displacement of striatal radioactivity for assessment of intrasynaptic dopamine. We will assess the feasibility of this paradigm for detecting l-dopa effects on the SPECT signal in subjects with PD with disease duration of greater than 4yrs and with a stable response to L-dopa. Each subject will undergo three [123I]-IBZM studies separated by 1-2 weeks. Subjects will be off medication for at least 12 h prior to study For each of the three scan days patients will receive a constant intravenous infusion of [123I]-IBZM over 4-5 hours to establish an equilibrium binding condition of the radiotracer at striatal D2/D3 receptors. Three baseline SPECT acquisitions will be obtained prior to medication dosing to establish a stable baseline. At approximately 5 h after the initiation of the infusion subjects will receive a single oral dose of either carbidopa/levodopa (37.5mg/150mg or 50mg/250mg), or carbidopa/levodopa/entacapone (either 37.5mg/150mg/200mg- STALEVO or 50/250mg/200mg).

ELIGIBILITY:
Main inclusion criteria:

* The patient is aged 30 years or older.
* Written informed consent is obtained.
* Patients have a diagnosis of idiopathic Parkinson's disease.
* Hoehn and Yahr stages for patients are I-III.
* Patients have a diagnosis> 4 yrs prior to screening
* Patients are treated with carbidopa/levodopa with > 300 mg levodopa.

Main exclusion criteria:

* The patient has atypical or drug-induced Parkinson's disease.
* The patient has dementia (MMSE 24).
* The patient has a clinically significant clinical laboratory values, and/or medical or psychiatric illness.
* The patient has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
* The patient has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* The patient has been treated with a dopamine agonist within the past 30 days.
* Concomitant treatment with Monoamine Oxidase (MAO)-inhibitors (except selegiline <10 mg/day) within 30 days prior to the screening visit
* Patient has a history of iodine allergy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-03; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the reduction from baseline in IBZM striatal uptake during a 6-8 hour assessment period after treatment. | 6-8hrs

SECONDARY OUTCOMES:
Secondary Measures include: Putamen and caudate uptake over time, UPDRS scores, and Pharmacokinetic analysis. | 6-8hrs

CONTACTS AND LOCATIONS:
Overall Officials: John P Seibyl, MD, Principal Investigator — Molecular NeuroImaging

REFERENCES:
- [Background] Castner SA, al-Tikriti MS, Baldwin RM, Seibyl JP, Innis RB, Goldman-Rakic PS. Behavioral changes and [123I]IBZM equilibrium SPECT measurement of amphetamine-induced dopamine release in rhesus monkeys exposed to subchronic amphetamine. Neuropsychopharmacology. 2000 Jan;22(1):4-13. doi: 10.1016/S0893-133X(99)00080-9. PMID 10633485
- [Background] de la Fuente-Fernandez R, Lu JQ, Sossi V, Jivan S, Schulzer M, Holden JE, Lee CS, Ruth TJ, Calne DB, Stoessl AJ. Biochemical variations in the synaptic level of dopamine precede motor fluctuations in Parkinson's disease: PET evidence of increased dopamine turnover. Ann Neurol. 2001 Mar;49(3):298-303. doi: 10.1002/ana.65.abs. PMID 11261503
- [Background] Laruelle M, D'Souza CD, Baldwin RM, Abi-Dargham A, Kanes SJ, Fingado CL, Seibyl JP, Zoghbi SS, Bowers MB, Jatlow P, Charney DS, Innis RB. Imaging D2 receptor occupancy by endogenous dopamine in humans. Neuropsychopharmacology. 1997 Sep;17(3):162-74. doi: 10.1016/S0893-133X(97)00043-2. PMID 9272483
- [Background] Seibyl JP, Woods SW, Zoghbi SS, Baldwin RM, Dey HM, Goddard AW, Zea-Ponce Y, Zubal G, Germine M, Smith EO, et al. Dynamic SPECT imaging of dopamine D2 receptors in human subjects with iodine-123-IBZM. J Nucl Med. 1992 Nov;33(11):1964-71. PMID 1432157
- [Background] Seibyl JP, Zea-Ponce Y, Brenner L, Baldwin RM, Krystal JH, Offord SJ, Mochoviak S, Charney DS, Hoffer PB, Innis RB. Continuous intravenous infusion of iodine-123-IBZM for SPECT determination of human brain dopamine receptor occupancy by antipsychotic agent RWJ-37796. J Nucl Med. 1996 Jan;37(1):11-5. PMID 8543979